CLINICAL TRIAL: NCT01186848
Title: Comparison of Fractional Photothermolysis Alone Versus Fractional Photothermolysis Plus Intense Focused Ultrasound for Treatment of Striae Distensae: A Prospective Randomized Control Trial.
Brief Title: Fractional Laser and Ultrasound for Striae Distensae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology - Head and Neck Surgery and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU34376
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Stretch Marks
Keywords: Stretch marks; Striae distensae
MeSH Terms: conditions — Striae Distensae

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1550-nm erbium-doped fractionated laser (Active Comparator)
  Interventions: Device: 1550-nm erbium-doped fractionated laser
- Combination treatment (Active Comparator): "micro-focused ultrasound" and "1550nm-fractionated laser"
  Interventions: Device: Combination treatment

INTERVENTIONS:
Device: Combination treatment — The contralateral side received the combination of micro-focused ultrasound treatment and 1550nm-fractionated laser alternatively every 2 weeks for a total of 4 treatments with site-match control area of baseline striae on each side.
  Arms: Combination treatment
Device: 1550-nm erbium-doped fractionated laser — Each side of thigh (or abdomen) was randomized to receive 1550nm-fractionated laser treatment every 2 weeks for a total of 4 treatments on one side.
  Arms: 1550-nm erbium-doped fractionated laser

SUMMARY:
This was a prospective randomized controlled study comparing the efficacy of micro-focused ultrasound when used in conjunction with 1550-nm erbium-doped fractionated laser versus 1550-nm erbium-doped fractionated laser alone for treatment of striae distensae(stretch marks).

Each side of thigh (or abdomen) was randomized to receive 1550nm-fractionated laser treatment every 2 weeks for a total of 4 treatments on one side and the contralateral side received micro-focused ultrasound treatment and 1550nm-fractionated laser alternatively every 2 weeks for a total of 4 treatments with site-match control area of baseline striae on each side.

The primary outcome measure by two dermatologists blindly compared the two areas of striae distensae on each side from live subjects using a questionnaire and quartile rating scale on the final follow-up visit.

This study was a pilot study designed to determine the feasibility of these procedures.

DETAILED DESCRIPTION:
The secondary outcomes were qualitative measurements of the mean striae width in the treatment area before(week0) and after treatment(week10) and subject satisfaction was determined by a satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years old male and female subjects with striae distensae on both thighs or both sides of the abdomen.
* Subjects are in good health.
* Subjects are willing, have the ability to understand and provide informed consent, and are able to communicate with the investigator.
* Subjects should be within a 20 lb range of their starting weight during in the study period.

Exclusion Criteria:

* Pregnant or lactating
* Subjects who are unable to understand the protocol or give informed consent.
* Subjects currently under treatment with corticosteroids for any medical problems or subjects who discontinued treatment less than 2 months prior to consent.
* Subjects who have had medical e.g usage of oral or topical retinoids, laser or surgical treatment for striae distensae within the last year.
* Subjects who have active skin disease or skin infection in the treatment area.
* Subjects who are allergic to lidocaine or prilocaine.
* Subjects who have a history of abnormal scarring.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period took place over approximately 6 months at an urban academic hospital.
Groups:
- Subjects Receiving Split Body Treatment: The unit of randomization was the individual side of a body within each subject to receive either 1550-nm erbium-doped fractionated laser treatment or the combination of the laser and ultrasound treatment for the treatment of striae.
  Each side of thigh (or abdomen) was randomized to receive 1550nm-fractionated laser treatment every 2 weeks for a total of 4 treatments on one side and the contralateral side received micro-focused ultrasound treatment and 1550nm-fractionated laser alternatively every 2 weeks for a total of 4 treatments with site-match control area of baseline striae on each side.
Period: Overall Study
Arm/Group | Subjects Receiving Split Body Treatment
Started | 30
Completed | 22
Not Completed | 8
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Receiving Split Body Treatment
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Live-rater by Two Blinded Dermatologists
Description: The primary outcome was a blinded rating of the treatment area (Fractional Laser vs. Fractional Laser plus Intense Focused Ultrasound) with the best cosmetic appearance. Two dermatologists blindly evaluated the treated and control areas of each side from live subjects on the final follow up visit (week 10). This was reported as percentages of participants for whom "1550-nm Erbium-doped Fractionated Laser" or "Micro-focused Ultrasound and 1550nm-fractionated Laser" resulted in the "best cosmetic appearance".
Time Frame: week 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- 1550-nm Erbium-doped Fractionated Laser: 1550-nm erbium-doped fractionated laser : Each side of thigh (or abdomen) was randomized to receive 1550nm-fractionated laser treatment every 2 weeks for a total of 4 treatments on one side.
- Combination Treatment: Combination of micro-focused ultrasound and 1550nm-fractionated laser : The treated sites were randomized to receive 1550nm-fractionated laser treatment every 2 weeks for a total of 4 treatments on one side and the contralateral side received micro-focused ultrasound treatment and 1550nm-fractionated laser alternatively every 2 weeks for a total of 4 treatments with site-match control area of baseline striae on each side.
Arm/Group | 1550-nm Erbium-doped Fractionated Laser | Combination Treatment
Number analyzed (Participants) | 22 | 22
Percentage of participants | 77.27 [54.63 to 92.18] | 22.73 [7.82 to 45.37]

ADVERSE EVENTS:
Arm/Group | 1550-nm Erbium-doped Fractionated Laser | Combination Treatment
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 1/30 | 3/30
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1550-nm Erbium-doped Fractionated Laser (N=30) | Combination Treatment (N=30)
pain (General disorders) | 0 (0) | 1 (1)
numbness (General disorders) | 0 (0) | 1 (1)
hyperpigmentation (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes